CLINICAL TRIAL: NCT02100098
Title: Peripheral Nerve Block Anaesthesia for Ankle Fracture Surgery - an Exploratory Study: Is Rebound Pain a Problem?
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Rune Sort, MD, Research Fellow, Herlev Hospital
Other Study IDs: PAnFractRebound-01
Record Dates: First submitted 2014-03-24; First posted 2014-03-31 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Postoperative Pain
Keywords: Ankle fracture; Nerve block; Postoperative pain; Pain profile; Rebound pain
MeSH Terms: conditions — Pain, Postoperative; Ankle Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this exploratory study is to characterize the postoperative pain profile of patients undergoing operation with internal fixation of an ankle fracture under nerve block anaesthesia. Special attention is payed towards the possible existence and clinical relevance of a rebound pain phenomenon upon cessation of the nerve block.

Results are used to guide the set up of a randomized controlled trial on the subject.

DETAILED DESCRIPTION:
Peripheral nerve blocks (PNB) are widely used as anaesthesia and postoperative pain control for surgery. Several studies have suggested multiple benefits of PNB's but primarily shown in elective surgery. Acute conditions like ankle fractures have a different pain profile and risks and benefits of PNB's have not been sufficiently researched in these cases.

A recent study (Goldstein et al. 2012) suggested that a rebound pain effect occur upon cessation of PNB effect defined as a pain increase to a significantly higher level than observed in patients with no PNB at the same point after surgery.

With this prospective, exploratory study we aim to examine the postoperative pain profile after PNB anaesthesia for ankle fracture surgery with focus on plausibility of a rebound pain effect (as defined above) upon PNB cessation.

Secondarily to explore a variety of factors related to postoperative pain profile and feasibility of PNB anaesthesia for ankle surgery including efficacy, risk factors, time factors as well as postoperative recovery and overall patient satisfaction. Results will provide focus for a following randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years old scheduled for internal fixation of an ankle fracture as defined above.
* Ability to read and understand Danish and give informed oral and written consent

Exclusion Criteria:

* Multitrauma patients / other simultaneous fractures
* Cognitive or psychiatric dysfunction causing expected inability to comply with study protocol
* "CAVE" nonsteroidal antiinflammatory drugs (NSAID) or Morphine or Local Anaesthetics as evaluated by anesthesiologist for any reason
* Primary investigator unavailable for PNB administration at scheduled time of operation
* Infection at PNB injection site
* Time from fracture to operation > 5 days
* Existing neuropathy with functional impairment of the fractured extremity
* Bodyweight < 50 kg
* Daily use of opioids > 2 weeks preoperatively
* Pregnancy
* Nephropathy requiring dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for internal fixation of an ankle fracture under PNB-anaesthesia at Herlev Hospital identified from the operation booking system via consecutive screening.
  Eligible ankle fractures will be those of anatomically uni-, bi- or trimalleolar composition including syndesmotic injury with distal but not proximal fibular fracture. The "third malleolus" is the distal posterior edge of the tibia. Fractures needing external fixation or causing ankle dislocation in need of imminent surgery is not eligible.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Clinically relevant pain increase based on analysis of Numeric Rating Scale pain score (NRS) area under the curve (AUC) for the time period 12-24 hours compared to 0-12 hours postoperatively. | 0, 2, 4, 6, 9, 12, 15, 18, 21 and 24 hours postoperatively
  Pain scores are assessed and marked by the patient on a 0-10 numeric rating pain scale (NRS).

SECONDARY OUTCOMES:
Opioid use 12-24 hours compared to 0-12 hours postoperatively | 0-24 hours continuous measurement
  Rescue morphine doses are administered intravenously via a patient controlled analgesia (PCA) pump when needed. Times of use are electronically registered.
Calculated Composite Score for the time intervals 0-24h, 0-12h and 12-24h postoperatively | 0-24 hours postoperatively
  We will calculate the "Silverman" composite score of opioid use and pain score combined. This in order to illustrate any increase in pain and to use for sample size calculations for a future randomised study on the subject.
Time to first opioid dose postoperatively | 0-24 hours postoperatively
Time to patient estimated cessation of block effect | 0-24 hours postoperatively
NRS day 1-7 as both "average" and "worst" of the day | Days 1-7 postoperatively
  NRS are filled out by the patient in a diary.
Daily opioid consumption day 1-7 | Days 1-7 postoperatively
  Registered in a diary.

OTHER OUTCOMES:
Clinically relevant pain increase based on analysis of Numeric Rating Scale pain score (NRS) area under the curve (AUC) after cessation of nerve block compared to before cessation of nerve block. | 0, 2, 4, 6, 9, 12, 15, 18, 21 and 24 hours postoperatively
  The average postoperative time to cessation of nerve block defining the time periods for this comparison will be defined after visual evaluation of the given pain profiles.
Score of the Quality of Recovery-15 (QoR-15) questionnaire preoperatively and on postoperative day 1. | Preoperatively and postoperative day 1
  Validation of the Danish translation of QoR-15 in this population of patients undergoing acute orthopaedic surgery under PNB-anaesthesia.
  A Danish version of the QoR-15 questionnaire is currently being validated in a mixed surgical patient population receiving surgery under general anaesthesia. We will attempt to validate the questionnaire on patients receiving nerve block (PNB) anaesthesia.
QoR-15 questionnaire score on day 1, 2 and 7 postoperatively | Postoperative day 1, 2 and 7.
Length of postoperative stay in hospital | Up to 3 weeks
Time to first meal/appetite postoperatively | 0-24 hours postoperatively
Incidence of postoperative nerve symptoms (PONS) on day 7 | Postoperative day 7
  Telephone interview
Postoperative nausea and vomiting (PONV) 24 hours postoperatively | 0-24 hours postoperatively
Antiemetic medication 24h postoperatively | 0-24 hours postoperatively
Time used for PNB administration | Preoperatively
Time to PNB effect on sensory and motor function | Preoperatively
Length of stay in the Operation Room (OR) - total and pre- and post-operatively | Operation day
Duration of surgery | Operation day
Partial block rate and Failed block rate | Operation day
  Partial = need for supplemental block preoperatively (if PNB seems insufficient after 30 min). Failed = need for General Anaesthesia.
Need for PACU admission postoperatively | Operation day
  Most patients are expected to be send directly to the Orthopaedic ward following surgery. If not, the reason is noted.

CONTACTS AND LOCATIONS:
Overall Officials: Rune Sort, MD, Principal Investigator — Department of Anaesthesiology, Herlev Hospital; Ann M Møller, Prof., DMSc, Study Director — Department of Anaesthesiology, Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Denmark, Denmark

REFERENCES:
- [Derived] Sort R, Brorson S, Gogenur I, Nielsen JK, Moller AM. Rebound pain following peripheral nerve block anaesthesia in acute ankle fracture surgery: An exploratory pilot study. Acta Anaesthesiol Scand. 2019 Mar;63(3):396-402. doi: 10.1111/aas.13290. Epub 2018 Nov 8. PMID 30411313